CLINICAL TRIAL: NCT01689350
Title: Prospective Study Based on Genetic Polymorphisms Related to Individual Variations of Side Effects of Cyclophosphamide in Systemic Lupus Erythematosus Treatment
Brief Title: A Prospective Study of Cyclophosphamide in Systemic Lupus Erythematosus Treatment
Acronym: SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lingyan Chen, Master Graduate Student, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012ZX09506001-004
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Cyclophosphamide; genotype-based therapy; prospective study
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): The cases in control group received traditional therapy that the initial dose of cyclophosphamide (CPA) was 0.2-0.6g/week injection according to clinical experience.
- Experimental Group (Experimental): Genetic: Genotype Detection To Genotype cases in the experimental group and divide them into three groups, including extensive metaboliser (EM), intermediate metaboliser (IM) and poor metaboliser (PM),with initial dose of CPA as 0.2g, 0.4g and 0.6g per week by injection, respectively.
  Interventions: Genetic: Genotype Detection

INTERVENTIONS:
Genetic: Genotype Detection — To Genotype cases in the experimental group and divide them into three groups, including extensive metaboliser (EM), intermediate metaboliser (IM) and poor metaboliser (PM).
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to compare the genotype-based personal prescription of cyclophosphamide with the traditional prescription.

DETAILED DESCRIPTION:
Cyclophosphamide (CPA) has been one of the most successful therapies for severe Systemic lupus erythematosus (SLE). However, cyclophosphamide can cause severe side effects, including bone marrow suppression, infection, gastrointestinal reaction, hemorrhagic cystitis, and the etc. Significant variation in efficacy and toxicity of CPA has been observed. Since the development of applicable therapeutic drug monitoring (TDM) of cyclophosphamide has been reported, it will help to improve the efficacy and reduce toxicities in SLE treatment. However, the TDM is a passive strategy which usually lags behind the appearance of toxicities. Therefore，it is especially crucial to give individuals genotype-based personal prescription of cyclophosphamide in order to gain the most effective therapies. Thus, the purpose of this study is to compare the genotype-based personal prescription of cyclophosphamide with the traditional prescription, in order to verify the efficacy of the genotype-based personal prescription.

ELIGIBILITY:
Inclusion Criteria:

* The American College of Rheumatology established eleven criteria in 1982,which were revised in 1997 as a classificatory instrument to operationalise the definition of SLE in clinical trials.

  1. Malar rash (rash on cheeks).
  2. Discoid rash (red, scaly patches on skin that cause scarring).
  3. Serositis: Pleurisy (inflammation of the membrane around the lungs) or pericarditis (inflammation of the membrane around the heart).
  4. Oral ulcers (includes oral or nasopharyngeal ulcers).
  5. Arthritis: nonerosive arthritis of two or more peripheral joints, with tenderness, swelling, or effusion.
  6. Photosensitivity (exposure to ultraviolet light causes rash, or other symptoms of SLE flareups).
  7. Blood-hematologic disorder-hemolytic anemia (low red blood cell count) or leukopenia (white blood cell count<4000/µl), lymphopenia (<1500/µl) or thrombocytopenia (<100000/µl) in the absence of offending drug. Hypocomplementemia is also seen, due to either consumption of C3 and C4 by immune complex-induced inflammation or to congenitally complement deficiency, which may predispose to SLE.
  8. Renal disorder: More than 0.5 g per day protein in urine or cellular casts seen in urine under a microscope.
  9. Antinuclear antibody test positive.
  10. Immunologic disorder: Positive anti-Smith, anti-ds DNA, antiphospholipid antibody, and/or false positive serological test for syphilis. Presence of anti-ss DNA in 70% of cases (though also positive with rheumatic disease and healthy persons).
  11. Neurologic disorder: Seizures or psychosis. For the purpose of identifying patients for clinical studies, a person has SLE if any 4 out of 11 symptoms are present simultaneously or serially on two separate occasions. In the meantime, the case has one of the following conditions or more;

  <!-- -->

  1. HIV (-);
  2. Signed the informed consent;
  3. Taking contraceptive measures during treatment period.

Exclusion Criteria:

* Poor compliance;
* With lupus mental damage complication, occurrence of epilepsy or unable to express subjective symptoms during the observation period.
* Taking drugs that affect cytochrome P450 2B6, cytochrome P450 3A4 and cytochrome P450 2C19, except corticosteroids.
* Abnormal liver function.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huang Min, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- School of Pharmaceutical Sciences Sun Yat-sen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: Cyclophosphamide (CPA) medication was according to the genotypes of SLE patients.
- Control Group: Cyclophosphamide (CPA) medication was according to the traditional experiences.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 47 | 45
Completed | 47 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: SLE patients who met the ACR criteria and applied CPA medication were included.
Groups:
- Control Group: 45 cases in control group received traditional therapy that the initial dose of cyclophosphamide (CPA) was 0.2-0.6g/week injection according to clinical experience.
- Experimental Group: 47 cases in experimental group were genotyped as extensive metaboliser (EM), intermediate metaboliser (IM) and poor metaboliser (PM）with initial dose of CPA as 0.2g, 0.4g and 0.6g per week by injection, respectively.
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.40 (13.28) | 31.15 (13.21) | 30.78 (13.17)
Sex/Gender, Customized [Number; unit: participants]
  Female | 38 | 40 | 78
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese Han | 45 | 47 | 92
Region of Enrollment [Number; unit: participants]
  China | 45 | 47 | 92
SLE patients [Number; unit: participants] | 45 | 47 | 92

OUTCOME MEASURES:

1. Primary Outcome: Adverse Reaction (Leucopenia)
Description: The count of white cells < 4.0 × 10ˆ9/L in SLE patient who received CPA medication was considered as CPA-induced leucopenia.
Time Frame: one month
Measure: Number; unit: participants
Groups:
- Experimental Group: CPA medication was according to the genotypes of SLE patients.
- Control Group: CPA medication was according to the traditional experiences.
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 47 | 45
participants | 6 [1.76 to 14.14] | 19 [1.76 to 14.14]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Null hypothesis: there is no difference between the control group and experimental group in terms of frequency of leucopenia.(α=0.05） Chi-square test was applied to test the difference. The Chi-square value was 10.08 and the P-value was 0.0015, which indicated that the null hypothesis could be rejected; Test type: Superiority or Other; p < 0.01, Chi-squared; Odds Ratio (OR) = 4.99, 95% CI 2-sided [1.76 to 14.14]

2. Secondary Outcome: Adverse Reaction ( Infection )
Description: Flu-like symptoms, Upper respiratory tract infection，and the etc.
Time Frame: one month
Measure: Number; unit: participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 47 | 45
participants | 8 | 16
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.01 to 7.13]

ADVERSE EVENTS:
Time Frame: One month for all the adverse events reporting.
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 6/47 | 19/45
Other Adverse Events (participants affected / at risk) | 8/47 | 16/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=47) | Control Group (N=45)
Leucopenia (Blood and lymphatic system disorders) | 6 | 19
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=47) | Control Group (N=45)
Infection (Infections and infestations) | 8 | 16

LIMITATIONS AND CAVEATS:
The sample size is too small to evaluate the significance of the cyclophosphamide (CPA) medication based on genotypes. We need to enroll more SLE patients in the following study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less